CLINICAL TRIAL: NCT06772662
Title: One Up, One Down: Analyzing Patient Preference on Cryotherapy Machine Tubing Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2410125
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Cryotherapy Tubing Placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tubing up (Active Comparator): Patients in this arm will have their cryotherapy machine tubing placed in the upwards position facing towards the head.
  Interventions: Procedure: Tubing Direction
- Tubing Down (Active Comparator): Patients in this arm will have their cryotherapy machine tubing placed in the downwards position facing towards the feet.
  Interventions: Procedure: Tubing Direction

INTERVENTIONS:
Procedure: Tubing Direction — We are studying the procedure of placing the Cryotherapy Tubing in two different directions: up vs down

SUMMARY:
The purpose of this research study is to better understand patient preference and their satisfaction rates with cryotherapy machines based on the direction of the tubing. This study will evaluate both satisfaction and pain of patients who use the cryotherapy machines in the two groups: tubing facing towards the head, and the other with tubing facing toward the feet.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an arthroscopic ACL reconstruction (CPT 29888) or MPFL reconstruction/augmentation with internal brace (CPT 27422 or 27429)
* Ages 10-18 years old at the time of surgery
* Patients who have access to a cryotherapy unit at the time of surgery

Exclusion Criteria:

* No ACL reconstruction (CPT 29888) nor MPFL reconstruction/augmentation with internal brace (CPT 27422 or 27429) performed during knee arthroscopy (i.e., isolated meniscus repair, synovectomy/debridement, etc.)
* Patients do not have access to a cryotherapy unit
* Patients less than 10 or older than 18 at the time of surgery

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Patients will prefer one direction of tubing placement over the other (up or down) by the end of 7 days post-op | 7 days
  Patients will report their opinion and preference of tubing placement based on the group they are randomized to at the end of 7 days post-op.

CONTACTS AND LOCATIONS:
Overall Officials: John Schlechter, DO, Principal Investigator — Children's Hospital of Orange County
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Age, Gender, Group Assignment, Outcome measures (satisfaction rates, pain scores).